CLINICAL TRIAL: NCT02557555
Title: Effects of Antenatal and Perinatal Education of Labor Analgesia Options on Maternal Anxiety, Labor Analgesia and Maternal Satisfaction With Labor Analgesia
Brief Title: Patient Education on Labor Analgesia Options
Status: Completed | Type: Observational
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Antonio Gonzalez Fiol, Anesthesiology Department, Assistant Professor Director of Obstetric Anesthesia Department of Anesthesiology, Rutgers, The State University of New Jersey
Other Study IDs: 20150001531
Record Dates: First submitted 2015-09-18; First posted 2015-09-23 (Estimated); Results first posted 2017-07-02 (Actual); Last update posted 2019-10-07 (Actual); Status verified 2019-10

CONDITIONS: Labor Analgesia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: educational information — patients will receive pamphlet on labor analgesia options.

SUMMARY:
The purpose of this study is to learn how the investigators can better educate pregnant patients about the options open to them for pain relief during labor. Patients will receive educational pamphlet during prenatal clinic visit and again on admission to labor and delivery. The options for analgesia will be discussed by anesthesia care provider. Patient will be asked to complete a survey on the post partum unit.

DETAILED DESCRIPTION:
Many analgesic options exist for laboring parturients, but labor may not be the best time to start informing patients of their options. Many patients begin the labor process with a plan in place for their analgesia. Unfortunately, internet resources regarding labor analgesia that are available to the lay parturient are poor and often lead to misconceptions about the options and their risks. A significant number of patients refuse neuraxial analgesia based on misunderstandings, concerns about the procedure, or a lack of faith in the provider. Some women want a "natural childbirth" and/or control over their labor experience. Our study aimed at providing information and alternatives for labor analgesia in a simple written format.

The investigators will provide information of available labor analgesia options (epidural, combined spinal/epidural, spinal, remifentanil patient-controlled analgesia, and intravenous opioids) to expecting mothers. Using a pamphlet written in English or Spanish disseminated to pregnant women in clinic and upon arrival in the labor and delivery unit, the procedures and their risks and benefits will be explained in simple terms. In the Labor and Delivery Unit the patients will have an opportunity to ask questions of the anesthesia care giver regarding the options for analgesia. After delivery while on F Green, patients will be asked to complete a questionnaire addressing their thoughts about the pamphlets and their overall satisfaction with their labor analgesia. The analysis will focus on the utility and effect of education materials on maternal informed consent for labor analgesia, on maternal choice of analgesia modality, and on maternal anxiety regarding their labor analgesia plan.

ELIGIBILITY:
Inclusion Criteria:

* Postpartum women ages 18 and older
* Patients who speak and read English or Spanish
* Patients who received our informational pamphlet while pregnant or in labor
* Patients who are able to consent and make medical decisions
* Patients undergoing labor or trial of labor after cesarean delivery
* Patients who undergo cesarean delivery after trial of labor

Exclusion Criteria:

* Patients unable or unwilling to complete questionnaire
* Patients unable to consent or make medical decisions
* Patients less than 18 years of age
* Patients unable to read and speak English or Spanish
* Patients in whom any of the analgesic options were contraindicated
* Patients with a history of an anxiety disorder
* Patients with precipitous labor or late presentation that precluded an analgesic intervention
* Patients with fetal distress that precluded an analgesic intervention
* Patients planned for elective cesarean section.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: pregnant females in prenatal clinic and labor suite
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Gonzalez-Fiol, MD, Principal Investigator — Rutgers, NJMS
Locations (1):
- University Hospital, Newark, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Labor Pain Control Pamphlet: All English or Spanish speaking patients were provided with a pamphlet during their prenatal visits and then again when entering the labor and delivery floor. The pamphlet contained information regarding labor analgesia alternatives (i.e Epidural, remifentanil patient controlled analgesia, morphine bolus, etc). After delivery, the patients were approached and asked to respond to a brief questionnaire.
Period: Overall Study
Arm/Group | Labor Pain Control Pamphlet
Started | 100
Completed | 100
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Labor Pain Control Pamphlet: All English or Spanish speaking patients were provided with a pamphlet during their prenatal visits and then again when entering the labor and delivery floor. The pamphlet contained information regarding labor analgesia alternatives (i.e Epidural, remifentanil PCA, morphine bolus, etc). After delivery, the patients were approached and asked to respond to a brief questionnaire.
Arm/Group | Labor Pain Control Pamphlet
Number analyzed (Participants) | 100
Age, Customized [Count of Participants; unit: Participants] — Patients age 18-45 admitted to labor and delivery
  Participants
    18-45 years | 100
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 100
Patients completing survey [Count of Participants; unit: Participants] | 100

OUTCOME MEASURES:

1. Primary Outcome: Survey to Determine Utility and Effect of Educational Materials
Description: In order to assess the educational value of the pamphlet provided to parturients we evaluated all the questions pertaining education. There is no nominal value reported in units as all the data is merely described as the percentage of patients responding to educational questions. For example, 93% of patients (91/98) responded Yes to the question -Do you think the pamphlet you received did a better job explaining your options for control of labor pain than what you answered in the previous question <patient research>?
Time Frame: expected average of no later than 48 hours following delivery
Population: The answers from 100 female patients, ages 18-45 admitted to the L&D who answered our survey were analyzed to gage the educational value of our labor analgesia informational pamphlet.
Measure: Number; unit: percentage of patients responding
Groups:
- Yes %: Percentage of patients responding Yes to one of the key questions of the study regarding education value of the pamphlet and anxiety level.
- No %: Percentage of patients responding no to the key questions regarding the provided pamphlet educational value or anxiety
Arm/Group | Yes % | No %
Number analyzed (Participants) | 100 | 100
percentage of patients responding
  Researched options for labor pain | 79 | 21
  Pamphlet better explained options for pain | 93 | 7
  Pamphlet should be given before onset labor pain | 97 | 3
  Pamphlet information helped to reduce anxiety | 90 | 10
  Information corrected any misconception: number analyzed (Participants) | 55 | 22
  Information corrected any misconception | 71 | 29
  Written information should always be available | 100 | 0
Statistical Analysis 1: Comparison: Yes % vs No %; Test type: Other — P-values corresponding to a test of equal proportions (yes/no- 50%/50%); p < 0.0001, Test of equal proportion (50/50) — Researched options for labor pain
Statistical Analysis 2: Comparison: Yes % vs No %; Test type: Other — P-values corresponding to a test of equal proportions (yes/no- 50%/50%); p < 0.0001, Test of equal proportion (50/50) — Pamphlet better explained options for pain
Statistical Analysis 3: Comparison: Yes % vs No %; Test type: Other; p < 0.0001, Test of equal proportion (50/50) — Pamphlet should be given before onset labor pain
Statistical Analysis 4: Comparison: Yes % vs No %; Test type: Other; p < 0.0001, Test of equal proportion (50/50) — Pamphlet information helped to reduce anxiety
Statistical Analysis 5: Comparison: Yes % vs No %; Test type: Other; p = 0.0002, Test of equal proportion (50/50) — Information corrected any misconception
Statistical Analysis 6: Comparison: Yes % vs No %; Test type: Other; p < 0.0001, Test of equal proportion (50/50) — Written information should always be available

ADVERSE EVENTS:
Time Frame: 1 year
Description: Given that the patients were asked to fill up a 24 question survey, no patient was exposed to any risk. That is, there was no interventional or placebo/drug arm in this study.
Arm/Group | Labor Pain Control Pamphlet
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2015-04-30): https://cdn.clinicaltrials.gov/large-docs/55/NCT02557555/Prot_000.pdf
  • Informed Consent Form (2015-04-30): https://cdn.clinicaltrials.gov/large-docs/55/NCT02557555/ICF_001.pdf
  • Statistical Analysis Plan (2018-10-31): https://cdn.clinicaltrials.gov/large-docs/55/NCT02557555/SAP_002.pdf